CLINICAL TRIAL: NCT06587490
Title: Total RadIoTherapy of Oligometastatic caNcerS (TRITONS)
Brief Title: Total RadIoTherapy of Oligometastatic caNcerS
Acronym: TRITONS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tyler Seibert, Radiation Oncologist, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 810616
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Oligometastatic Malignant Solid Neoplasm
Keywords: Stereotactic ablative radiotherapy; oligometastatic cancer; randomized phase III trial; biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SABR+SOC (Experimental): stereotactic ablative radiotherapy (SABR) plus standard of care (SOC) cancer therapy
  Interventions: Radiation: stereotactic ablative radiotherapy
- SOC (No Intervention): standard of care (SOC) cancer therapy

INTERVENTIONS:
Radiation: stereotactic ablative radiotherapy — Stereotactic ablative radiotherapy is a highly focused radiation treatment that gives an intense dose of radiation concentrated on a tumor, while limiting the dose to the surrounding organs.
  Other Names: SABR
  Arms: SABR+SOC

SUMMARY:
This is a Phase III non-blinded randomized study evaluating patients with oligometastatic cancers (up to 10 metastases). Subjects are randomized 1:1 to stereotactic ablative radiotherapy (SABR) plus standard of care therapies versus standard of care therapies alone. The investigators will measure progression-free survival at 2 years based on the hypothesis that subjects treated with SABR plus standard of care will not experience disease progression for a longer period of time than subjects treated with standard of care alone. The investigators will also measure overall survival and safety of SABR, as well as biomarkers that may help predict, in the future, who will benefit from the SABR treatment.

DETAILED DESCRIPTION:
Patients with metastatic solid malignancies are generally deemed incurable. Systemic therapies (cytotoxic chemotherapy, immunotherapy, hormonal therapy, etc.) can be effective for prolonging life, but cancers will eventually become resistant, prompting transition to second-line therapies that are often more toxic and/or more expensive with diminishing oncologic benefit. In patients with relatively few detectable metastases, SABR to visible tumors may substantially delay progression and thus improve quality of life. Unfortunately, most patients with metastatic disease will eventually die from their cancer. Stereotactic ablative radiotherapy (SABR) is highly effective, often achieving long-term local control. Previous studies demonstrated that SABR improves survival and quality of life in patients with oligometastatic cancer. However, these studies were small and not randomized. Thus, this randomized study will better evaluate the efficacy and safety of SABR in oligometastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Age at least 18 years.
4. Deemed eligible to undergo standard systemic therapy and SABR to metastatic sites (i.e., patient has adequate health and life expectancy, and treatment is not contraindicated).
5. Histopathologic confirmation of a solid malignancy.
6. Newly diagnosed or progressive metastasis (at least 1 and no more than 10 discrete distant metastases visible on staging imaging. At least one metastatic lesion must be outside the brain parenchyma) for which a new line of systemic therapy is started or resumed.
7. New systemic therapy for metastatic disease initiated no more than 6 months prior to randomization.
8. For participants able to become pregnant: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during active SABR treatment.
9. For participants able to cause a pregnancy: use of condoms or other methods to ensure effective contraception with partner during active SABR treatment.

Exclusion Criteria:

1. Pregnancy.
2. Contraindications to radiotherapy, including interstitial lung disease if thoracic radiation is planned; Crohn's disease if the gastrointestinal tract will receive radiotherapy; active connective tissue disorders such as scleroderma or uncontrolled lupus; moderate or severe liver dysfunction (Child Pugh B or C) if the patient has liver metastases.
3. Prior radiation therapy to an area requiring treatment in the present study, if the composite dose would exceed normal tissue constraints specified by UC San Diego Radiotherapy Standards and Guidelines (published by the Department of Radiation Medicine and Applied Sciences), or by local institutional radiotherapy dose constraints for safety and efficacy.
4. Malignant pleural effusion or malignant ascites.
5. Leptomeningeal disease in the central nervous system.
6. Metastatic disease in a site where it is not possible to safely treat with SABR to the doses specified in the trial.
7. Any unresected metastasis >5 cm in largest diameter or >3 cm in the brain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2033-11 (Estimated); Study Completion 2034-11 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  Rate of Progression Free Survival in the two study arms

SECONDARY OUTCOMES:
All-grade and grade ≥3 toxicity | 2 years
  All-grade and grade ≥3 toxicity per CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Seibert, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No